CLINICAL TRIAL: NCT03939962
Title: Phase Ⅱ Study of PD-1 Inhibitor Combined With FOLFOX Neoadjuvant Therapy for Resectable Gastric and Gastroesophageal Junctional Adenocarcinoma
Brief Title: Camrelizumab Combined With FOLFOX Neoadjuvant Therapy for Resectable Gastric and Gastroesophageal Junctional Adenocarcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HNGC-004
Record Dates: First submitted 2019-05-04; First posted 2019-05-07 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2021-05

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Folfox protocol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): Neoadjuvant therapy:SHR1210 combined with FOLFOX repeat every 14 days for a total of 4 cycles.
  Adjuvant therapy:SHR1210 combined with chemotherapy (the specific regimen will be chosen at the discretion of the investigator), every 14 days for a total of 4 cycles. After that, the patients will receive camrelizumab monotherapy for up to 1 year (from the first SHR1210 treatment).
  Interventions: Drug: SHR1210 combined with FOLFOX

INTERVENTIONS:
Drug: SHR1210 combined with FOLFOX — 1. SHR1210, iv, 200 mg d1, 30-minute intravenous infusion, repeated every 14 days.
  2. FOLFOX: Oxaliplatin 85mg/m2 ivgtt 2h d1; 5-fluorouracil 400mg/m2 iv d1; leucovorin 400mg/m2 ivgtt 2h d1,5-fluorouracil 2400mg/m2 CIV 46h, repeated every 14 days Patients who have no disease progression and can tolerate surgery receive surgery. When the investigator believes that the patient is not suitable for continued medication or according to the RECIST 1.1 standard, the evaluation is PD and the medication is over. The PD-1 monoclonal antibody does not allow for reductions and can only delay or suspend medication.

SUMMARY:
The aim of this study is to observe the efficacy, safety, postoperative pathological response rate and survival benefit of immume checkpoint inhibitor PD-1 SHR1210 combined with chemotherapy in neoadjuvant therapy of locally advanced resectable gastric and gastroesophageal junction adenocarcinoma. In addition ，the investigators will explore the relationship between the immunophenotype of gastric cancer and the efficacy and drug resistance of immunotherapy combined with chemotherapy, and screen out biomarkers that can predict the efficacy of immunotherapy.

DETAILED DESCRIPTION:
Neoadjuvant chemotherapy and neoadjuvant radiotherapy and chemotherapy can not only improve the surgical resection rate and postoperative pathological remission rate, but also prolong the postoperative recurrence-free survival and benefit patients.Recent studies have confirmed that immume point inhibitors PD-1 and CTLA-4 monoclonal antibody have a certain effect in advanced gastric and gastroesophageal junction adenocarcinoma which had experienced multi-line treatment. Furthermore，the FOLFOX protocol is recommended as a new adjuvant treatment for locally advanced gastric cancer.In order to further improve the surgical resection rate and survival rate by improving the efficacy of neoadjuvant therapy for locally advanced gastric and gastroesophageal junction adenocarcinoma, the investigators selected PD-1 monoclonal antibody combined with FOLFOX neoadjuvant therapy for locally advanced gastric and gastroesophageal junctions Adenocarcinoma.The aim of this study is to observe the efficacy, safety, postoperative pathological response rate and survival benefit of immume checkpoint inhibitor PD-1 SHR1210 combined with chemotherapy in neoadjuvant therapy of locally advanced resectable gastric and gastroesophageal junction adenocarcinoma. In addition ，the investigators will explore the relationship between the immunophenotype of gastric cancer and the efficacy and drug resistance of immunotherapy combined with chemotherapy, and screen out biomarkers that can predict the efficacy of immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. 18-73 years old; male or female
2. confirmed gastric and gastroesophageal junction adenocarcinoma by Gastroscopic biopsy histopathological examination
3. Imaging (CT/MRI) and ultrasound gastroscopy confirmed: cT ≥ T2 and / or regional lymph node positive (N +);
4. ECOG score: 0~2 points;
5. Expected survival period ≥ 12 weeks;
6. A histological specimen can be provided for secondary testing;
7. The main organ function meets the following criteria within 7 days before treatment:

   Blood routine examination criteria (without blood transfusion within 14 days):

   Hemoglobin (HB) ≥ 90g / L; The absolute value of neutrophils (ANC) ≥ 1.5 × 109 / L; Platelet (PLT) ≥ 80 × 109 / L (2) Biochemical examinations must meet the following criteria: Total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal (ULN); Alanine aminotransferase (ALT) Aspartate aminotransferase (AST) ≤ 2.5 * ULN; serum creatinine (Cr) ≤ 1.5 * ULN or creatinine clearance (CCr) ≥ 60ml / min; (3) Doppler ultrasound assessment: left ventricular ejection fraction (LVEF) ≥ normal low limit (50%).
8. Women of childbearing age should agree to use contraceptives (such as intrauterine devices, contraceptives or condoms) during the study period and within 6 months after the end of the study; negative serum or urine pregnancy test within 7 days prior to study enrollment and must be non-lactating patients; men should agree to patients who must use contraception during the study period and within 6 months after the end of the study period.
9. The patient volunteered to participate in the study and signed an informed consent form;

Exclusion Criteria:

1. Exceeding or currently suffering from other malignant tumors within 5 years, except for cervical cancer in situ, non-melanoma skin cancer and superficial bladder tumors [Ta (non-invasive tumor), Tis (in situ carcinoma) And T1 (tumor infiltrating basement membrane)];
2. Patients with a high risk of bleeding or fistula due to the apparent invasion of adjacent organs (aorta or trachea);
3. Before starting treatment， subject administrated corticosteroids (day> 10 mg equivalent dose prednisone), or other immunosuppressive drugs for systemic treatment of a disease within 14 days . In the absence of active autoimmune disease, >10 mg of daily prednisone equivalent dose of inhaled or topical steroid and adrenal replacement steroid doses are permitted;
4. Anyone who has received any anti-tumor treatment in the past;
5. Significantly malnourished patients. Exclusion is performed if the patient is receiving intravenous fluids or is required to be hospitalized for continuous infusion therapy. Patients with good nutrition control ≥ 28 days can be enrolled before randomization;
6. Participants who received live/attenuated vaccine within 30 days of the first treatment;
7. Unresolved toxicity due to any previous treatment above CTC AE4.0 Level 2, excluding neurotoxicity of ≤2 caused by hair loss and oxaliplatin;
8. Allergic reactions and adverse drug reactions:

   1. a history of allergies to the ingredients of the study drug;
   2. contraindications to any study drug (fluorouracil or oxaliplatin) in the chemotherapy regimen.
9. Patients with any severe and/or uncontrolled disease, including:

   1. patients with hypertension who are not well controlled by antihypertensive drug (systolic blood pressure ≥150 mmHg, diastolic blood pressure ≥100 mmHg);
   2. with grade I or higher myocardial ischemia or myocardial infarction, arrhythmia (including QTc ≥ 480ms) and ≥ grade 2 congestive heart failure (New York Heart Association (NYHA) classification);
   3. Severe or uncontrolled disease or active infection (≥CTCAE grade 2 infection), which the investigator believes may increase the risk associated with study participation, study drug administration, or affect the subject's ability to receive study medication;
   4. Renal failure requires hemodialysis or peritoneal dialysis;
   5. a history of immunodeficiency, including HIV-positive or other acquired, congenital immunodeficiency disease, or a history of organ transplantation;
   6. Patients with diabetes who have poor glycemic control (fasting blood glucose (FBG) > 10 mmol/L); subjects with active, known or suspected autoimmune diseases. Subjects with type 1 diabetes, residual hypothyroidism caused by autoimmune thyroiditis requiring hormone replacement therapy, and skin diseases that do not require systemic treatment (such as vitiligo, psoriasis or alopecia) can be enrolled;
   7. patients with seizures and requiring treatment;
   8. The subject has an interstitial lung disease that is symptomatic or may interfere with the discovery or management of suspected drug-related lung toxicity; previous and current subjects with a history of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-associated pneumonia, severe impaired lung function, etc. that may interfere with the detection and management of suspected drug-related lung toxicity;
10. Patients with gastrointestinal diseases such as intestinal obstruction (including incomplete intestinal obstruction) or those who may have caused gastrointestinal bleeding, perforation or obstruction;
11. Patients who underwent surgical treatment, incisional biopsy or significant traumatic injury within 28 days prior to enrollment;
12. In the 4 weeks prior to enrollment, patients with any bleeding event ≥ CTCAE 3 have unhealed wounds, ulcers or fractures;
13. Overactive/venous thrombosis events within 3 months, such as cerebrovascular accidents (including transient ischemic attacks), deep static Pulmonary thrombosis and pulmonary embolism;
14. Prepare or accept previous allogeneic or allogeneic bone marrow transplantation, including liver transplantation;
15. According to the investigator's judgment, there is a concomitant disease that seriously harms the patient's safety or affects the patient's completion of the study;
16. Cannot perform biopsy to provide histological specimens;
17. those who have a history of psychotropic substance abuse and are unable to quit or have a mental disorder; Prepare or accept previous allogeneic or allogeneic bone marrow transplants, including liver transplants;
18. Urine routine showed urinary protein ≥ 2+ and confirmed 24-hour urine protein quantitation > 1.0 g;
19. Patients with brain metastases;
20. Patients who have participated in other clinical trials of anti-tumor drugs within four weeks.

Ages: 18 Years to 73 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-07-24 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
R0 resection rate | Up to approximately 16 weeks
  The percentage of patients who have no residual cancer cells (gross or microscopically) at the resection margins.
pathological complete response (pCR) rate | Up to approximately 16 weeks
  The percentage of patients with no residual cancer cells at the primary cancer site and N(-) per histological evaluation.

SECONDARY OUTCOMES:
Near pathological complete response (near-pCR) rate | Up to approximately 16 weeks
  Near-pCR rate is defined as the percentage of patients with grade 0-1 tumors per NCCN tumor regression grading (TRG).
Overall survival(OS) | From randomization to the date of death (up to approximately 4 years)
  OS is defined as the time from the first dose to all-cause death.
Progression-free survival(PFS) | up to 2 years
  PFS is defined as the time from the first dose to objective disease progression or death.
Disease-free survival (DFS) | From randomization to the date of recurrence or death (up to approximately 4 years)
  DFS is defined as the time from the postoperative baseline imaging evaluation to disease recurrence or death in subjects who are disease-free after surgery.
Percentage of Participants Who Experience One or More Adverse Events (AEs) | up to approximately 1 years
  The incidence and grade of adverse events (including serious adverse events and immune-related adverse events) will be determined per NCI-CTCAE 4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Liu, Principal Investigator — Henan Cancer Hospital/The affiliated Cancer Hospital of ZhengZhou university
Locations (1):
- Henan Cancer Hospital/The affiliated Cancer Hospital of ZhengZhou university, Zhengzhou, Henan, China

REFERENCES:
- [Derived] Zhao Y, Li D, Zhuang J, Li Z, Xia Q, Li Z, Yu J, Wang J, Zhang Y, Li K, Xu S, Li S, Ma P, Cao Y, Liu C, Xu C, Liu Z, Wei J, Zhang C, Qiao L, Gao X, Hou Z, Liu C, Zheng R, Wang D, Liu Y. Comprehensive multi-omics analysis of resectable locally advanced gastric cancer: Assessing response to neoadjuvant camrelizumab and chemotherapy in a single-center, open-label, single-arm phase II trial. Clin Transl Med. 2024 May;14(5):e1674. doi: 10.1002/ctm2.1674. PMID 38685486